CLINICAL TRIAL: NCT02764411
Title: Onreltea (Brimonidine) Gel In Pediatric Patients With Capillary Malformations: A Prospective, Open-label, Cohort Study
Brief Title: Onreltea (Brimonidine) Gel In Pediatric Patients With Capillary Malformations
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor enrollment, lack of feasibility
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Elena Pope, Professor of Paediatrics, University of Toronto Fellowship Director and Section Head, Paediatric Dermatology., The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000051364
Record Dates: First submitted 2016-04-19; First posted 2016-05-06 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Capillary Malformations
Keywords: Capillary malformations; Onrealtea; port-wine stain; treatment; topical
MeSH Terms: conditions — Capillary Malformations, Congenital, 1; Port-Wine Stain | interventions — Brimonidine Tartrate; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Onreltea ( Brimonidine) (Experimental): All the patients enrolled in the study will apply Onreltea ( Brimonidine 0.33%) gel on the affected skin area for 12 weeks (from Day 0 to Week 12 visit).
  Interventions: Drug: Brimonidine 0.33% gel

INTERVENTIONS:
Drug: Brimonidine 0.33% gel — Topical application of Brimonidine 0.33% gel on Capillary Malformation (CM) lesion once daily for 12 weeks
  Other Names: Onreltea

SUMMARY:
Capillary Malformations (CM) affect a significant proportion of otherwise healthy children and may lead to psychological discomfort if left untreated. A significant proportion of untreated lesions undergo soft tissue thickening and darker discoloration later in life due to progressive ectasia of the affected vessels. While laser treatment is available, its use may be limited due to need for repeated sedation/general anesthetic use, partial response and cost.

The investigators propose to conduct an open-label, prospective, cohort study using Onreltea ( Brimonidine) gel for treatment of facial capillary malformations in children. The study medication will be applied topically on affected area of the skin daily for 12 weeks. Follow up visits will occur at at Week 1,4,8,12, and 16 to assess the efficacy and safety of the proposed treatment.

The study second aim is to explore the feasibility of conducting a multicenter placebo controlled study.

DETAILED DESCRIPTION:
The investigators are planning to enroll in the study 20 participants at SickKids.

It is a prospective, open label, cohort study. Patients enrolled in the study will be followed at the Hospital For Sick Children for 16 weeks. They will come for the study visits 6 times: in 1 week, 4,8,12, and 16 weeks after the treatment has been started. During each study visit the study investigators will assess any changes in the characteristics of CM lesion(s) captured by a Chromometer *, Analogue Scale and Erythema Assessment tools. Participants or their parents will assess the changes at the final study visit (VAS and EA tools).

Patients will be provided with study medication for all duration of the study treatment (12 weeks).

The results of the treatment will be compared with the baseline data to evaluate the efficacy and safety of Onreltea (Brimonidine) gel in children with facial capillary malformations.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of facial capillary malformation (port-wine stain, PWS) made by a dermatologist
* age: 12-17 years of age
* weight > 45 kg
* lesions with a surface area < 100 cm2
* signed consent and assent for study participation

Exclusion Criteria:

* skin breakdown overlying the malformation due to other dermatological conditions (e.g. eczema, psoriasis)
* current or treatment with laser the past 3 months
* other topical treatments used within the past 4 weeks (e.g. rapamycin, corticosteroids, calcineurin inhibitors, etc)
* known chronic renal or hepatic disorders
* known cardiovascular disorders
* other systemic medications that potentially interact with Brimonidine (opiates, chlorpromazine, methyphenidate, reserpine, etc)
* mixed capillary/ venous or lymphatic malformations
* known allergy to one of the constituents of Onreltea
* pregnancy, or sexually active subjects of child-bearing potential (CBP), unwilling to use contraception during the study (such as barrier method, or oral contraceptives).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The change in the color of the capillary malformation using Chroma meter values (Δa, ΔE) at 12 weeks. | 12 weeks
  Measurement of erythema will be performed using Chroma Meter, CR-400, Konica, Minolta, Osaka, Japan. The meter readings will result in 3 values: L- refers to the relative light intensity, ranging from 0 (black) to +100 (white); a-captures color saturation, ranging from +60 (green) to -60 (red) and b- captures color spectrum from +60 (blue) to -60 (yellow). In most studies both, changes in a (Δa) and overall changes in the composite score (ΔE calculated as √((ΔL*before-ΔL*after)^2+(Δa*before-Δa*after)^2+(Δb*before-ΔL*after)^2 ) are obtained.

SECONDARY OUTCOMES:
Changes in the color of the lesion (Δa, ΔE) at each follow up visit including the last visit at 16 weeks compared to baseline | 1,4,8,16 weeks
  Same as in primary outcome measure
Changes in CEA scores at 12, 16 weeks compared to baseline | 12 and 16 weeks
  A Clinician Erythema Assessment scale (CEA), consisting of a 0-4 numerical scale as follows:
  0- clear skin, no erythema
  1. almost clear skin, slight redness
  2. mild erythema, definite redness
  3. moderate erythema, marked redness
  4. severe erythema, fiery redness
Changes in the iVAS at 12 and 16 weeks compared to baseline | 12 and 16 weeks
  Investigator's assessment of changes on the Visual Analogue Scale ( iVAS)
Correlation between iVAS, pVAS, CEA, pEA and Chroma Meter values | 1,4,8,12,16 weeks
  pVAS - patient/parent's Visual Analogue Scale assessment; pEA- patient/parent Erythema Assessment
Percentage of patients achieving 75% and 100% resolution of the lesion | 12 weeks
  by iVAS and chromo meter values
Frequency of observed and reported adverse events (AE) | 16 weeks
  AE documented in patient diary and mentioned at each study visit

OTHER OUTCOMES:
Predictors for a good response, defined as at least 50 % change in the erythema measured using Chroma Meter (a* after compared to a* before) at 12 weeks mark | 12 weeks
  Predictors for a good response, defined as at least 50 % change in the erythema measured using Chroma Meter (a* after compared to a* before) at 12 weeks mark. Percent of participants with predictors for a good response.
Percentage difference in Chroma Meter values (L -relative light intensity, a - color saturation, b - color spectrum) between treated and untreated lesions (control) | 1,4,8,12 and 16 weeks
  Changes in value ( e.g. "a") between baseline and Week *, calculated in % for investigational lesion, minus changes in value "a" between baseline and Week * , calculated in % for the control lesion.
  (a (inv.Week*) - a (inv. Baseline)/ a (inv. Baseline)) x 100% -- (a (contr. Week*) - a (contr. Baseline)/ a ( contr. baseline)) x 100%
Percentage of patients experiencing flare-up (defined as reoccurrence of the red discoloration) at the end of the study (16 weeks) | 16 weeks
  Percentage of patients experiencing flare-up (defined as reoccurrence of the red discoloration) at the end of the study (16 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pope, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital For Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No